CLINICAL TRIAL: NCT03679091
Title: Low-dose of Ticagrelor and Standard-dose Clopidogrel on Platelet Effects in Chinese Patients With Stable Coronary Artery Disease: a Randomized, Single-blind, Crossover Clinical Study
Brief Title: Low-dose of Ticagrelor and Standard-dose Clopidogrel on Platelet Effects in Chinese Patients With Stable CAD.
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: First Affiliated Hospital of Harbin Medical University (Other)
Responsible Party: Principal Investigator, Yue LI, Professor, First Affiliated Hospital of Harbin Medical University
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: CHD-201845
Record Dates: First submitted 2018-09-04; First posted 2018-09-20 (Actual); Last update posted 2021-12-21 (Actual); Status verified 2021-12

CONDITIONS: Platelet Reactivity
Keywords: Ticagrelor; clopidogrel; coronary artery disease; platelet reactivity
MeSH Terms: conditions — Coronary Artery Disease | interventions — Ticagrelor; Clopidogrel

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- low-dose ticagrelor (Experimental): To observe the safety and efficacy of low-dose ticagrelor in Chinese patients with Stable Coronary Artery Disease
  Interventions: Drug: low-dose ticagrelor; Drug: Clopidogrel
- clopidogrel (Active Comparator): To observe the safety and efficacy between low-dose ticagrelor and standard-dose clopidogrel.
  Interventions: Drug: low-dose ticagrelor; Drug: Clopidogrel

INTERVENTIONS:
Drug: low-dose ticagrelor — low-dose ticagrelor (60.0 mg once daily) for 7 days,followed by a 2-week washout period then a 7 days crossover phase of clopidogrel (75mg once daily).
Drug: Clopidogrel — clopidogrel (75mg once daily) for 7 days,followed by a 2-week washout period then a 7 days crossover phase of low-dose ticagrelor (60.0 mg once daily).

SUMMARY:
Ticagrelor has been demonstrated to provide a more rapid and more powerful inhibition of platelet aggregation compared with clopidogrel in coronary artery disease (CAD) patients. However, current guidelines recommend ticagrelor 90 mg twice daily might not be suitable for patients of Chinese. Therefore, the investigators performed this study to observe the efficacy of 60-mg ticagrelor in comparison to 75-mg clopidogrel in Chinese patients with stable CAD.

DETAILED DESCRIPTION:
Dual antiplatelet therapy with aspirin and a P2Y12 receptor antagonist is the established standard of care in ACS patients. Although a popular P2Y12 receptor inhibitor, clopidogrel is not the most potent antiplatelet agent due to its metabolic activation. Metabolic activation of clopidogrel depends on multiple cytochrome P450 (CYP) enzymes, including CYP2C19, which can delay the onset of its activity; in addition, some populations carry a reduced-function allele of the CYP2C19 gene. Notably, poor drug metabolism of clopidogrel is more common in Asian populations compared with other international regions, due to the prevalence of CYP2C19 reduced-function alleles in these patients. A recent study indicated that Asians might have different adverse event profiles (thrombophilia and bleeding) and "therapeutic window" compared with white subjects, suggesting that regional differences may influence the altered response of clopidogrel to the onset of thrombotic events.

Ticagrelor is an orally administered, reversibly-binding, direct-acting P2Y12 receptor antagonist used clinically for the prevention of atherothrombotic events in patients with ACS. Guidelines give a recommendation on the use of dual antiplatelet therapy (DAPT) support ticagrelor 90 mg twice daily over clopidogrel 75 mg daily in addition to aspirin in ACS patients with or without ST-segment elevation. Increasing evidence indicated that Asian patients showed higher active metabolite exposure rates and stronger pharmacodynamic responses than their Caucasian subjects when treated with the same oral doses of prasugrel .In Korea and Japan, it has been reported that low doses of ticagrelor might have a more potent inhibition of platelet aggregation (IPA) than clopidogrel in healthy subjects and patients with stable coronary artery disease, respectively .In our previous study, the investigators found that half-dose ticagrelor produced similar inhibitory effects on platelet aggregation as standard-dose ticagrelor and exerted significantly stronger effects than clopidogrel in patients with ACS and one-quarter standard-dose ticagrelor provided greater degree of platelet inhibition than clopidogrel in patients with stable CAD. Furthermore, standard-dose ticagrelor (180mg loading dose [LD], then 90mg twice daily) has a significant increase in the risk of bleeding and incidence rate of dyspnea, and that higher discontinuation rates due to adverse effects compared to clopidogrel. A recent study demonstrated that maximum plasma concentration and area under the plasma concentration-time curve of ticagrelor (90 mg twice daily) and its active metabolite (AR-C124910XX) tended to be approximately 40% higher in healthy Chinese volunteers compared with Caucasian subjects. Notably, poor drug metabolism of clopidogrel is more common in Asian populations compared with other international regions, due to the prevalence of CYP2C19 reduced-function alleles. The data suggested that a low dose of ticagrelor might be more appropriate for Chinese patients.

The objectives of this study were to evaluate the effects of ticagrelor (60.0mg daily) in comparison to clopidogrel (75mg daily) on platelet reactivity in Chinese patients with stable CAD.

ELIGIBILITY:
Inclusion Criteria:

* Patients were eligible to participate if they were aged ≥18 years and ≤ 75 Years
* Subjects had documented stable CAD (defned as stable angina pectoris and objective evidence of CAD, a previous MI, or previous revascularization with percutaneous coronary intervention or coronary artery bypass grafting)
* Women were required to be postmenopausal or surgically sterile
* Patients who were taking clopidogrel or ticagrelor were required to discontinue these agents at least 14 days before randomization

Exclusion Criteria:

* Acute coronary syndrome (ACS)
* planned use of glycoprotein IIb/IIIa receptor inhibitors, adenosine diphosphate (ADP) receptor antagonists other than the study medication, or anticoagulant therapy during the study period
* platelet count <10*10^4/ul
* creatinine clearance rate < 30ml/min
* diagnosed as respiratory or circulatory instability (cardiac shock, severe congestive heart failure NYHA II-IV or left ventricular ejection fraction < 40%)
* a history of bleeding tendency
* allergy to aspirin, ticagrelor or clopidogrel
* diabetes patients

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2018-08-29 (Actual); Primary Completion 2019-02-28 (Actual); Study Completion 2019-02-28 (Actual)

PRIMARY OUTCOMES:
The platelet inhibition ratio. | up to 2 months
  Verifynow was used to measure platelet inhibition ratio.

SECONDARY OUTCOMES:
The platelet aggregation ratio. | up to 2 months
  Light transmission aggregometry method was used to measure platelet aggregation ratio.

CONTACTS AND LOCATIONS:
Overall Officials: Yue Li, professor, Principal Investigator — First Affiliated Hospital of Harbin Medical University
Locations (1):
- VerifyNow, Harbin, California, China